CLINICAL TRIAL: NCT06139523
Title: Optimize Pediatric OCT (Optical Coherence Tomography) Imaging: a Pilot Study
Brief Title: Optimize Pediatric OCT Imaging
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00113627
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Retinal Disease; Glaucoma; Optic Nerve Diseases
Keywords: Optical Coherence Tomography (OCT)
MeSH Terms: conditions — Retinal Diseases; Glaucoma; Optic Nerve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group 1: Healthy adult volunteers: Healthy adult volunteers recruited from the patient population, students or employees of Duke University or Duke Eye Center (n=10)
  Interventions: Device: Investigational contact OCT system; Device: Investigational noncontact OCT system:
- Pediatric participants: Pediatric patients with eye disease recruited from the patient population of Duke Eye Center (n=20)
  Interventions: Device: Investigational contact OCT system; Device: Investigational noncontact OCT system:

INTERVENTIONS:
Device: Investigational contact OCT system — Theia imaging is developing handheld OCT systems bring state of the art OCT to the infant bedside. The Theia 1 widefield imaging system is a light weight, high speed (300 kHz), wide field of view (110°) OCT system that address the limitations of current commercial OCT systems. The system is cart mounted, enabling portable, bedside imaging. The system uses a 300 kHz swept source laser operating in 1060nm regime. The Theia system follows the same safety standards as all applicable laser safety standards (ANSI z80.36 or ISO 15004) as the currently approved prior OCT devices. This nearly 10-fold increase in acquisition speed dramatically reduces imaging time and enables acquisition of full retinal volumes in infants. The 110° field of view is provided via a re-usable contact lens that can be sterilized between imaging sessions.
  Other Names: Theia 1 widefield imaging system
Device: Investigational noncontact OCT system: — The investigational noncontact handheld OCT systems in this study is developed at Duke University as the result of collaboration between the Departments of Ophthalmology (Cynthia Toth, MD) and Biomedical Engineering (Joseph Izatt, PhD). This investigational device was previously reviewed and approved for use in adults, children, and neonates in nursery by:
  * Intraoperative OCT Guidance of Intraocular Surgery study's (Pro00016827) Data Safety and Monitoring Board Plus (DSMB+) (PI: Toth and Izatt)
  * The Analyzing Retinal Microanatomy in Retinopathy of Prematurity to Improve Care study (Pro00069721) Data Safety and Monitoring Committee (DSMC) (PI: Toth) The systems were declared non-significant risk by the Duke University Health System (DUHS) Institutional Review Board under Pro00016827. Staff from the DUHS Clinical Engineering Department evaluated the systems and found that they meet the accepted hospital standards for electrical safety.
  Other Names: Ultracompact swept source OCT system

SUMMARY:
Handheld optical coherence tomography (OCT) has become an important imaging modality to evaluate the pediatric retina. The objective of this pilot study is to compare a new contact OCT system (Theia Imaging) with an investigational noncontact OCT system (Duke Biomedical Engineering) to assess their ability to image the pediatric retina.

The investigators hypothesize that the contact OCT system is superior in imaging larger areas of the retina (larger field-of-view), while it has similar resolution to image the retina substructures (non-inferior image quality).

DETAILED DESCRIPTION:
Handheld optical coherence tomography (OCT) has become an important imaging modality to evaluate the pediatric retina. The objective of this pilot study is to compare a new contact OCT system (Theia Imaging) with an investigational noncontact OCT system (Duke Biomedical Engineering) to assess their ability to image the pediatric retina.

The investigators plan to enroll 10 healthy adult volunteers and 20 pediatric patients in clinic or undergoing examination under anesthesia. This is an observational study. There are no known risks associated with handheld OCT imaging and no adverse events identified imaging with our prior investigational imaging with the same system. There is a risk of corneal abrasion with the contact imaging system (Theia imaging), however, this system is used in the setting of other contact imaging systems (such as RetCam fundus photography).

Imaging data will be downloaded to a secure server for protocol image processing, segmentation, and analysis per protocol in the Duke Advanced Research in SD/SSOCT Imaging (DARSI) Laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 - Healthy adult volunteers
* Subject is able and willing to consent to study participation
* Subject is more than 18 years of age
* Healthy adult volunteers without known ocular issues other than refractive error
* Pregnancy Reasonably Excluded Guide (PREG) evaluation on women of childbearing potential
* Group 2 - Pediatric participants
* Health care provider, knowledgeable of protocol, agrees that study personnel could contact the parent/legal guardian
* Parent/legal guardian is able and willing to consent to study participation
* Pediatric patient less than 18 years of age in Duke Eye Center ophthalmology clinics or undergoing clinically-indicated examination under anesthesia at Duke Eye Center

Exclusion Criteria:

* Group 1 - Healthy adult volunteers
* Students or employees under direct supervision of the investigators
* Subjects with prior problems with pupil dilation
* Pregnant woman if receiving dilating drops
* Group 2 - Pediatric participants
* Parent/legal guardian unwilling or unable to provide consent
* Participant has a health or eye condition that preclude eye examination or retinal imaging (such as corneal opacity or cataract)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Group 1 - Healthy adult volunteers (n=10). Participants over the age of 18 without known ocular issues other than refractive error.
  Group 2 - Pediatric participants (n=10). Participants under the age of 18 being seen at Duke Eye Center for ocular abnormailities.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Presence of abnormal retinal microanatomy as measured by OCT reading | Single imaging session (day 1)
Severity of abnormal retinal microanatomy as measured by OCT reading | Single imaging session (day 1)
Retinal thickness at the fovea and surrounding optic nerve as measured by OCT analysis | Single imaging session (day 1)
  Retinal thickness (microns) at the fovea and surrounding optic nerve.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott AW, Farsiu S, Enyedi LB, Wallace DK, Toth CA. Imaging the infant retina with a hand-held spectral-domain optical coherence tomography device. Am J Ophthalmol. 2009 Feb;147(2):364-373.e2. doi: 10.1016/j.ajo.2008.08.010. Epub 2008 Oct 9. PMID 18848317
- [Background] Chavala SH, Farsiu S, Maldonado R, Wallace DK, Freedman SF, Toth CA. Insights into advanced retinopathy of prematurity using handheld spectral domain optical coherence tomography imaging. Ophthalmology. 2009 Dec;116(12):2448-56. doi: 10.1016/j.ophtha.2009.06.003. Epub 2009 Sep 18. PMID 19766317
- [Background] Maldonado RS, Izatt JA, Sarin N, Wallace DK, Freedman S, Cotten CM, Toth CA. Optimizing hand-held spectral domain optical coherence tomography imaging for neonates, infants, and children. Invest Ophthalmol Vis Sci. 2010 May;51(5):2678-85. doi: 10.1167/iovs.09-4403. Epub 2010 Jan 13. PMID 20071674
- [Background] Maldonado RS, Freedman SF, Cotten CM, Ferranti JM, Toth CA. Reversible retinal edema in an infant with neonatal hemochromatosis and liver failure. J AAPOS. 2011 Feb;15(1):91-3. doi: 10.1016/j.jaapos.2010.11.016. PMID 21397814
- [Background] Maldonado RS, O'Connell R, Ascher SB, Sarin N, Freedman SF, Wallace DK, Chiu SJ, Farsiu S, Cotten M, Toth CA. Spectral-domain optical coherence tomographic assessment of severity of cystoid macular edema in retinopathy of prematurity. Arch Ophthalmol. 2012 May;130(5):569-78. doi: 10.1001/archopthalmol.2011.1846. PMID 22232366
- [Background] Chen X, Mangalesh S, Dandridge A, Tran-Viet D, Wallace DK, Freedman SF, Toth CA. Spectral-Domain OCT Findings of Retinal Vascular-Avascular Junction in Infants with Retinopathy of Prematurity. Ophthalmol Retina. 2018 Sep;2(9):963-971. doi: 10.1016/j.oret.2018.02.001. Epub 2018 Mar 21. PMID 30506013
- [Background] Chen X, Prakalapakorn SG, Freedman SF, Vajzovic L, Toth CA. Differentiating Retinal Detachment and Retinoschisis Using Handheld Optical Coherence Tomography in Stage 4 Retinopathy of Prematurity. JAMA Ophthalmol. 2020 Jan 1;138(1):81-85. doi: 10.1001/jamaophthalmol.2019.4796. PMID 31774474
- [Background] Mangalesh S, Bleicher ID, Chen X, Viehland C, LaRocca F, Izatt JA, Freedman SF, Hartnett ME, Toth CA. Three-dimensional pattern of extraretinal neovascular development in retinopathy of prematurity. Graefes Arch Clin Exp Ophthalmol. 2019 Apr;257(4):677-688. doi: 10.1007/s00417-019-04274-6. Epub 2019 Feb 21. PMID 30790072
- [Background] Mangalesh S, Sarin N, McGeehan B, Prakalapakorn SG, Tran-Viet D, Cotten CM, Freedman SF, Maguire MG, Toth CA; BabySTEPS Group. Preterm Infant Stress During Handheld Optical Coherence Tomography vs Binocular Indirect Ophthalmoscopy Examination for Retinopathy of Prematurity. JAMA Ophthalmol. 2021 May 1;139(5):567-574. doi: 10.1001/jamaophthalmol.2021.0377. PMID 33792625